CLINICAL TRIAL: NCT05154344
Title: Real World Effectiveness of Capmatinib in Patients With Advanced MET-dysregulated NSCLC Included in the French Compassionate Use Program (ATU)
Brief Title: RW Effectiveness of Capmatinib in Advanced MET-dysregulated NSCLC Included in the French Compassionate Use Program (ATU)
Acronym: CapmATU
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-2104
Record Dates: First submitted 2021-11-02; First posted 2021-12-13 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: MET Alterations; Non Small Cell Lung Cancer; METex14 Mutations
Keywords: Expanded access program; Capmatinib; MET TKIs; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capmatinib — Available through expanded access
  Other Names: Tabrecta

SUMMARY:
CapmATU study will evaluate time to treatment failure, progression-free survival, overall survival, best response and safety in patients with advanced MET-dysregulated non-small cell lung cancer who received capmatinib as part of an expanded access program. Those outcomes will be correlated to clinical, pathological, and radiological characteristics of patients.

DETAILED DESCRIPTION:
Capmatinib has been approved in the USA and Japan. In France, a compassionate use for capmatinib has been approved in June 2019 for patients with MET alterations, including METex14 mutations and MET amplification. In March 2021, 204 patients are or have been treated with compassionate use capmatinib as part of this program, most of them (n=175) harboring a METex14 mutation.

So far, data on activity and safety of new-generation MET TKIs are still sparse and only based on prospective clinical studies. The CapmATU study is a unique opportunity to describe patients' characteristics and outcomes, and confirm effectiveness of capmatinib in a large cohort of METex14 NSCLC. Moreover, it will provide original real-world evidence (RWE). RWE can be used in oncology to further characterize the safety and efficacy of drugs in the post-marketing setting. This may include confirmation of clinical benefit for regulatory purposes, expansion of labeling claims to new indications, testing of alternate doses and schedules of drugs, and assessment of drug activity in biomarker-defined subgroups and other special populations. This may be even more important in the context of METex14 NSCLC patients since no real world data with new generation MET TKIs have been reported so far. Indeed, this study will allow to determine whether the antitumor activity of capmatinib reported in the GEOMETRY-MONO-1 study can be observed in less selected patients. Given the older age and associated comorbidities of METex14 NSCLC patients, most of them may not be eligible to a clinical trial, thus emphasizing the need for real-world evidence. Finally, the biological part of this study (CapmATU-BIO) will offer opportunity to identify biomarkers of sensitivity or acquired resistance to capmatinib, which is a poorly explored field of research so far.

In this context, the objectives of this non-interventional retrospective French population-base study are to describe the characteristics of patients with MET-dysregulated NSCLC, assess effectiveness and safety of capmatinib in these patients and identify biomarkers of benefit from capmatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced or metastatic NSCLC (Stage IIIB or IV accordingly to American Joint Committee on Cancer [AJCC] classification) at time of capmatinib initiation
* Presence of a MET dysregulation diagnosed on tumor sample and/or on liquid biopsy
* Patients who were informed about the study and accepted for their data to be collected.
* Patients who received at least one dose of treatment with capmatinib as part of the compassionate use program (ATU), whatever the line of treatment.
* Selection period spans from June 1st 2019 (date of start of French ATU) until August 31st 2021 for first dose of capmatinib.
* Age >18 y

Exclusion Criteria:

* Patients enrolled in a clinical trial assessing treatment with capmatinib. (ATU was granted to patients unable to meet eligibility criteria for on-going recruiting trials, unable to participate to other clinical trials, or because other medical interventions were not considered appropriate or acceptable).
* Patients who were included in the French Early Access Program (ATU program) but did not receive any capmatinib treatment.
* Patients who have expressed explicit refusal to collect his or her data
* Patients with a psychiatric history that hinders the comprehension of the information leaflet
* Patients under curatorship or guardianship
* Unability to obtain data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC harboring a METex14 mutation receiving capmatinib as part of the French compassionate use program (ATU).
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
time to treatment failure | 2 years
  time to treatment failure in patients with advanced NSCLC harboring a METex14 mutation receiving capmatinib as part of the French compassionate use program (ATU)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Lille
  - CHU, Tours